CLINICAL TRIAL: NCT04591210
Title: Evaluation of the Potential Benefit of Renin-angiotensin System Inhibitors (RASi, ACEi/ARB) in High-risk Patients With COVID-19. The COVID-RASi Trial
Brief Title: The COVID-RASi Trial (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTO-3212
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Cardiovascular Diseases
Keywords: cardiovascular risk factors; corona virus; COVID-19; severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); Angiotensin-converting enzyme inhibitors; ACEi; Renin-angiotensin system inhibitors; RASi; Angiotensin receptor blockers; ARB
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Treatment (Standard of Care) (No Intervention): Participants will be treated as per standardized care pathway according to province/state and institutional guidelines. Physicians will be reminded not to start ACEi or ARB throughout admission or to outpatients until active study participation is complete at 28 days post symptoms.
- ACEi treatment (Experimental): The physician will initiate any ACE inhibitor and dose at their discretion.
  Interventions: Drug: Angiotensin converting enzyme inhibitor
- ARB treatment (Experimental): The physician will initiate any ARB and dose at their discretion.
  Interventions: Drug: Angiotensin II Receptor Blockers

INTERVENTIONS:
Drug: Angiotensin converting enzyme inhibitor — The study recommends physicians to select an ACEi with proven benefit in cardiovascular diseases such as perindopril, ramipril or enalapril. Lab values will be obtained during baseline. The patient will be followed by the physician clinically, with recommended laboratory testing in one week, including renal function, potassium assessment, and dose adjustments as appropriate.
  Arms: ACEi treatment
Drug: Angiotensin II Receptor Blockers — The study recommends physicians to select evidence-based ARBs such as candesartan or valsartan or losartan. Lab values will be obtained during baseline. The patient will be followed by the physician clinically, with recommended laboratory testing in one week, and dose adjustments as appropriate.
  Arms: ARB treatment

SUMMARY:
The COVID-RASi study is an international randomized clinical trial that will evaluate the potential benefit of angiotensin modulators on clinical outcomes, in COVID-19 patients. The purpose of this study is to determine if renin-angiotensin system inhibitors (RASi), with angiotensin-converting enzyme inhibitors (ACEi) or angiotensin II receptor blockers (ARB), has a beneficial effect in patients with COVID-19 infections, by reducing ICU admission, ventilator requirement or death. We would also like to determine if there are differences between ACEi and ARB therapeutic treatments. With the increasing potential of long COVID symptoms, at the 1 year follow up, a primary endpoint will be the quality of life of study participants, as assessed by ongoing symptoms and/or the standardized questionnaires.

DETAILED DESCRIPTION:
The goal is to determine if RASi with ACEi or ARB, has a beneficial effect in patients with COVID-19 infections, by reducing hospitalizations, ICU admission, ventilator requirement or death.

This is a multi-centre study, conducted in major centres treating COVID-19 patients in-hospital and in various outpatient settings.

Patients admitted to hospital or outpatients that test positive for COVID-19 and meet the inclusion/exclusion criteria will be eligible to participate in this study. All study participants will not be on RASi (ACEi/ARB) treatment at the time of consent. Participants will be randomized to initiation of ACEi vs ARB treatment vs no RASi treatment as part of care for COVID-19 in a 1:1:1 ratio.

The patient will be followed by their physician according to usual clinical care. Sites will complete research-related follow-ups at 24 hours, 7 and 28 days to asssess patient's clinical status, side effects and the achievement of clinical endpoints by telephone interviews. Phone call follow ups will also be conducted at 6 months and 12 months after enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient with COVID-19 diagnosis with laboratory confirmation within the last 30 days AND
* Age 40 years old or greater if outpatient OR age 18 years old or greater if inpatient (admitted to the hospital) at time of recruitment

Exclusion Criteria:

* Contraindication to ARB or ACEi, including severe aortic stenosis and angioedema
* Patients who are currently on active treatment with ARB/ACEi
* Known bilateral renal artery stenosis
* Systolic BP ≤90 mmHg
* eGFR<30 ml/min, if not receiving dialysis treatment
* K>5.5 mmol/L on screening laboratory testing
* Recent history of dizziness, vertigo, related to hypotension or orthostatic hypotension, that can lead to contraindication to ACEI/ARBs
* Acute respiratory distress syndrome requiring invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Death | 28 days
  Within first 28 days post randomization
Mechanical ventilation | 28 days
  Within first 28 days post randomization
ICU admission | 28 days
  Within first 28 days post randomization
Major Adverse Cardiac Events (MACE) | 28 days
  Within first 28 days post randomization
Hospitalizations | 28 days
  Within first 28 days post randomization
Quality of life of study participants | 1 year
  Assessed by ongoing symptoms and standardized questionnaires, scale to assess overall health 1-100, 100 is the best, higher score means better outcome
Quality of life of study participants | 1 year
  Assessed by ongoing symptoms and standardized questionnaires- scale to assess overall health 1-100, 100 is the best, higher score means better outcome

SECONDARY OUTCOMES:
Days alive and out of hospital | 30 days
Days alive and out of hospital | 180 days
Cardiovascular mortality | 1 year
All cause hospitalization | 1 year
Percent of patients require intensive care | 1 year
Percent of patients requiring ventilation | 1 year
Percent of patients requiring dialysis | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Liu, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (31):
- Brazil (21):
  - Centro de Pesquisa Clinicas Dr Marco Mota, Maceió, Alagoas
  - Centro de Pesquisas em Diabetes e Doencas Endocrino-Metabolicas, Fortaleza, Ceará
  - Santa Casa de Itabuna, Itabuna, Estado de Bahia
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Clinica da Unimed Campo Grande, Campo Grande, Minas Gerais
  - Clinica de Campo Grande, Campo Grande, Minas Gerais
  - Nucleo de Pesquisa Clinica SS, Curitiba, Paraná
  - Hospital Agamenom Magalhaes, Recife, Pernambuco
  - Pronto Socorro Cardiologico de Pernambuco Recife, Recife, Pernambuco
  - Hospital Eduardo Campos da Pessoa Idosa, Estância, Recife
  - Instituto Atena de Pesquisa Clinica, Natal, Rio Grande do Norte
  - Hospital Universitar Canoas, Canoas, Rio Grande do Sul
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Universitario Sao Francisco na Providencia de Deus, Bragança Paulista, São Paulo
  - Instituto de Pesquisa Clinica de Campinas, Campinas, São Paulo
  - Hospital Bela Vista, Consolação, São Paulo
  - Hospital de Julho, São Paulo, São Paulo
  - Instituto de Coracao, São Paulo, São Paulo
  - Instituto Prevent Senior, São Paulo, São Paulo
  - Instituto Goiano de Oncologia e Hematologia, Goiânia
- Canada (2):
  - Alberta Health Services, Edmonton, Alberta
  - University of Ottawa Heart Institute, Ottawa, Ontario
- Mexico (8):
  - Hospital de Infectologia Dr Daniel Mendez Fernandez, Azcapotzalco, Mexico City
  - Hospital General de Zona 20, La Margarita, Puebla
  - Hospital General Regional No 2, El Marqués, Querétaro
  - Unidad de Medicina Familiar No 77, Ecatepec de Morelos, State of Mexico
  - Hospital General zona 11, Xalapa, Veracruz
  - Unidad de Medicina Familiar No 10, Xalapa, Veracruz
  - Hospital General 1, IMSS, Mexico City
  - Hospital General de zona 27- IMSS, Mexico City

IPD SHARING:
Plan to Share IPD: No